CLINICAL TRIAL: NCT02970305
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Pimavanserin as Adjunctive Treatment for the Negative Symptoms of Schizophrenia
Brief Title: Efficacy and Safety of Pimavanserin as Adjunctive Treatment for the Negative Symptoms of Schizophrenia (ADVANCE)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ACADIA Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACP-103-038; 2016-003436-20 (EudraCT Number)
Record Dates: First submitted 2016-11-18; First posted 2016-11-22 (Estimated); Results first posted 2020-12-22 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — pimavanserin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pimavanserin (Experimental): Drug- pimavanserin 34 mg, 20 mg, or 10 mg taken as two tablets + background antipsychotic, once daily by mouth
  Interventions: Drug: Pimavanserin
- Placebo (Placebo Comparator): Placebo, taken as two tablets + background antipsychotic, once daily by mouth
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pimavanserin — Pimavanserin 34 mg, 20 mg, or 10 mg, taken as two tablets, once daily by mouth
  Arms: Pimavanserin
Drug: Placebo — Placebo, taken as two tablets, once daily by mouth
  Arms: Placebo

SUMMARY:
To evaluate the efficacy and safety of adjunctive pimavanserin compared with adjunctive placebo in the treatment of the negative symptoms of schizophrenia

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients, between 18 and 55 years of age
2. A clinical diagnosis of schizophrenia with a minimum duration of 1 year
3. Has predominant negative symptoms according to predefined study criteria
4. The main background antipsychotic with which the subject is being treated must be one of the antipsychotics listed below:

   * Aripiprazole
   * Aripiprazole long-acting injectables:

     * Abilify Maintena®
     * Aristada®
   * Risperidone
   * Risperidone long-acting injection
   * Olanzapine
   * Lurasidone
   * Cariprazine
   * Brexpiprazole
   * Asenapine

Exclusion Criteria:

1. Patient has a psychiatric disorder other than schizophrenia
2. A urine drug screen (UDS) result at Baseline that indicates the presence of any tested prohibited substance of potential abuse, except marijuana

   a. Patients with a result indicating the presence of marijuana are permitted if they agree to abstain from marijuana use during the study and the medical monitor approves the subject's participation
3. Patient has current evidence of a serious and/or unstable psychiatric, neurologic, cardiovascular, respiratory, gastrointestinal, renal, hepatic, hematologic, or other medical disorder, including cancer or malignancies, which would affect the patient's ability to participate in the program
4. Patient has had a myocardial infarction in the last six months
5. Patient has a family or personal history or symptoms of long QT syndrome
6. Patient has been hospitalized due to inadequate family support or care at the patient's primary residence, during the 8 weeks prior to screening

Patients will be evaluated at screening to ensure that all criteria for study participation are met. Patients may be excluded from the study based on these assessments (and specifically if it is determined that their baseline health and psychiatric condition do not meet all pre-specified entry criteria).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 403 (Actual)
Dates: Start 2016-11-04 (Actual); Primary Completion 2019-10-16 (Actual); Study Completion 2019-10-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (81):
- United States (30):
  - Phoenix, Arizona
  - Rogers, Arkansas
  - Bellflower, California
  - Lemon Grove, California
  - Norwalk, California
  - San Diego, California
  - Santa Ana, California
  - Torrance, California
  - Hialeah, Florida
  - Lauderhill, Florida
  - Miami, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Decatur, Georgia
  - Marietta, Georgia
  - Chicago, Illinois
  - Hoffman Estates, Illinois
  - Wichita, Kansas
  - Ann Arbor, Michigan
  - Las Vegas, Nevada
  - Berlin, New Jersey
  - Albuquerque, New Mexico
  - Rochester, New York
  - Charlotte, North Carolina
  - Durham, North Carolina
  - Oklahoma City, Oklahoma
  - Downingtown, Pennsylvania
  - Charleston, South Carolina
  - Irving, Texas
  - Richardson, Texas
- Bulgaria (5):
  - Plovdiv
  - Sofia
  - Targovishte
  - Tserova Koria
  - Varna
- Canada (4):
  - Penticton, British Columbia
  - Chatham, Ontario
  - Montreal, Quebec
  - Toronto
- Czechia (4):
  - Hradec Králové, Vekose
  - Pilsen
  - Prague
  - Říčany
- Hungary (6):
  - Kalocsa, Bács-Kiskun Megya
  - Budapest, Pest County
  - Budapest
  - Debrecen
  - Gyula
  - Pécs
- Poland (4):
  - Bialystok
  - Bydgoszcz
  - Lublin
  - Pruszcz Gdański
- Russia (8):
  - Roshchino, Leningradskaya Oblast'
  - Plekhanovo, Lipetsk Oblast
  - Saint Petersburg
  - Samara
  - Smolensk
  - Stavropol
  - Yaroslavl
  - Yekaterinburg
- Serbia (4):
  - Belgrade
  - Kovin
  - Kragujevac
  - Niš
- Spain (5):
  - Barcelona
  - Madrid
  - Oviedo
  - Valladolid
  - Zamora
- Ukraine (11):
  - Dnipro
  - Hlevakha
  - Kharkiv
  - Kherson
  - Kyiv
  - Lviv
  - Odesa
  - Oleksandrivka
  - Poltava
  - Smila
  - Vinnytsia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bugarski-Kirola D, Abbs B, Odetalla R, Liu IY, Darwish M, DeKarske D. Adherence to Background Antipsychotic and Pimavanserin in Patients with Schizophrenia: Post Hoc Analyses from the ENHANCE and ADVANCE Studies. Patient Prefer Adherence. 2024 Jan 19;18:207-216. doi: 10.2147/PPA.S436041. eCollection 2024. PMID 38264323
- [Derived] Darwish M, Bugarski-Kirola D, Passarell J, Owen J, Jaworowicz D, DeKarske D, Stankovic S. Pimavanserin Exposure-Response Analyses in Patients With Schizophrenia: Results From the Phase 2 ADVANCE Study. J Clin Psychopharmacol. 2022 Nov-Dec 01;42(6):544-551. doi: 10.1097/JCP.0000000000001611. Epub 2022 Oct 3. PMID 36190440
- [Derived] Bugarski-Kirola D, Arango C, Fava M, Nasrallah H, Liu IY, Abbs B, Stankovic S. Pimavanserin for negative symptoms of schizophrenia: results from the ADVANCE phase 2 randomised, placebo-controlled trial in North America and Europe. Lancet Psychiatry. 2022 Jan;9(1):46-58. doi: 10.1016/S2215-0366(21)00386-2. Epub 2021 Nov 30. PMID 34861170

RESULTS

PARTICIPANT FLOW:
Groups:
- Pimavanserin: Treatment was to be started at a daily dose of pimavanserin 20 mg; this dose was to be continued for the first 2 weeks of treatment . Subsequently, during the flexible-dosing period of double-blind treatment period (Weeks 2-8), the dose could be continued unchanged, increased to up to 34 mg daily, or decreased to up to 10 mg daily at the investigator's discretion, based on clinical benefit and safety/tolerability. No dose adjustments were allowed during the fixed-dosing period of the double-blind treatment period (Weeks 8-26).
  Patients were to continue their background antipsychotic treatment
- Placebo: Pimavanserin matching placebo once daily
  Patients were to continue their background antipsychotic treatment
Period: Overall Study
Arm/Group | Pimavanserin | Placebo
Started | 201 | 202
Completed | 172 | 174
Not Completed | 29 | 28
Not completed — Adverse Event | 10 | 6
Not completed — Lack of Efficacy | 1 | 1
Not completed — Noncompliance with study drug | 2 | 4
Not completed — Protocol Violation | 2 | 2
Not completed — Withdrawal by Subject | 12 | 11
Not completed — Not further specified | 1 | 2
Not completed — Lost to Follow-up | 1 | 2

BASELINE CHARACTERISTICS:
Population: Patients randomised and treated with at least one dose of study medication
Groups:
- Total: Total of all reporting groups
Arm/Group | Pimavanserin | Placebo | Total
Number analyzed (Participants) | 201 | 202 | 403
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.7 (9.37) | 36.7 (9.24) | 37.2 (9.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 65 | 135
  Male | 131 | 137 | 268
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 10 | 15 | 25
  White | 187 | 186 | 373
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Schizophrenia diagnosis confirmed by SCID-5-CT [Count of Participants; unit: Participants] — SCID-5-CT: Structured Clinical Interview for DSM-5, Clinical Trials Version
  Participants | 201 | 202 | 403

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 26 in the Negative Symptom Assessment-16 (NSA-16) Total Score
Description: The NSA-16 is a semi-structured interview and a validated scale containing 16 items for evaluating negative symptoms of schizophrenia, i.e. the reduction or absence of emotional expression and volitional behaviors normally present in a healthy person. Items are scored based on behaviors during the interview (items 1-4, 6, 7, 9, 11, 15, 16) or previous 7 days (items 5, 8, 10, 12-14) on a 6-point scale from 1 to 6. The NSA-16 total score is the sum of item scores. It can range from 16 to a maximum of 96, with higher scores denoting more severe negative symptoms in schizophrenia.
Time Frame: From baseline to Week 26
Population: Patients who were randomised and treated (received at least one dose of study drug) and had a baseline value and at least one post-baseline value for NSA-16 total score.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Pimavanserin | Placebo
Number analyzed (Participants) | 199 | 201
score on a scale
  Baseline | 61.8 (0.60) | 61.0 (0.61)
  Change from baseline to Week 26: number analyzed (Participants) | 174 | 173
  Change from baseline to Week 26 | -10.5 (0.69) | -8.8 (0.69)
Statistical Analysis 1: Comparison: Pimavanserin vs Placebo; Test type: Superiority; p = 0.0434, Mixed-effects model for repeated measure; Difference in MMRM LSMs = -1.9, 95% CI 2-sided [-3.8 to -0.1], Standard Error of Mean 0.95

2. Secondary Outcome: Change From Baseline to Week 26 in the Personal and Social Performance Scale (PSP) Score
Description: The PSP is a validated 100-point (1 to100) single-item rating scale to assess the psychosocial functioning of subjects with schizophrenia. Ratings are based on 4 main areas i.e. (a) socially useful activities, including work and study; (2) personal and social relationships, (3) self-care; and (4) disturbing and aggressive behaviors. The time period assessed is "past month". Higher scores denote better psychosocial functioning
Time Frame: From baseline to Week 26
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Pimavanserin | Placebo
Number analyzed (Participants) | 199 | 201
score on a scale
  Baseline | 47.2 (0.83) | 46.7 (0.76)
  Change from baseline to Week 26: number analyzed (Participants) | 174 | 173
  Change from baseline to Week 26 | 8.1 (0.70) | 8.4 (0.75)

3. Secondary Outcome: Proportion of Negative Symptom Assessment-16 (NSA-16) Responders at Week 26
Description: The NSA-16 is a semi-structured interview and a validated scale containing 16 items for evaluating negative symptoms of schizophrenia, i.e. the reduction or absence of emotional expression and volitional behaviors normally present in a healthy person. Items are scored based on behaviors during the interview (items 1-4, 6, 7, 9, 11, 15, 16) or previous 7 days (items 5, 8, 10, 12-14) on a 6-point scale from 1 to 6. The NSA-16 total score is the sum of item scores. It can range from 16 to a maximum of 96, with higher scores denoting more severe negative symptoms in schizophrenia.
  NSA-16 responders were defined as patients with at least 20, 30, 50, or 75% percentage improvement in NSA-16 total score from baseline.
Time Frame: From baseline to Week 26
Population: Patients who were randomised and treated (received at least one dose of study drug) and had a baseline value and at least one post-baseline value for NSA-16 total score and had no missing values at Week 26.
Measure: Count of Participants; unit: Participants
Arm/Group | Pimavanserin | Placebo
Number analyzed (Participants) | 174 | 173
Participants
  At least 20% improvement | 93 | 84
  At least 30% improvement | 56 | 51
  At least 50% improvement | 21 | 16
  At least 75% improvement | 4 | 2

4. Secondary Outcome: Change From Baseline to Week 26 in NSA-16 Global Negative Symptoms Rating
Description: The global negative symptoms rating of the NSA-16 assesses overall severity on a 7-point scale from 1 to 7, with higher scores denoting more severe negative symptoms in schizophrenia.
Time Frame: From baseline to Week 26
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Pimavanserin | Placebo
Number analyzed (Participants) | 199 | 201
score on a scale
  Baseline | 4.7 (0.05) | 4.8 (0.05)
  Change from baseline to Week 26: number analyzed (Participants) | 174 | 173
  Change from baseline to Week 26 | -0.7 (0.06) | -0.7 (0.06)

5. Secondary Outcome: Change From Baseline (CFB) to Week 26 in NSA-16 Domain Scores
Description: The NSA-16 is a semi-structured interview and a validated scale containing 16 items for evaluating negative symptoms of schizophrenia, i.e. the reduction or absence of emotional expression and volitional behaviors normally present in a healthy person. Items are scored based on behaviors during the interview (items 1-4, 6, 7, 9, 11, 15, 16) or previous 7 days (items 5, 8, 10, 12-14) on a 6-point scale from 1 to 6. The NSA-16 domain scores are the sum of item scores in each domain i.e. communication (min score 4, max score 24), emotion/affect (min 3, max 18), social involvement (min 3, max 18), motivation (min 4, max 24), and retardation (min 2, max 12); with higher scores denoting more severe negative symptoms in schizophrenia.
Time Frame: From baseline (BL) to Week 26
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Pimavanserin | Placebo
Number analyzed (Participants) | 199 | 201
score on a scale
  Communication, BL | 12.3 (0.22) | 12.3 (0.21)
  Communication, CFB to Week 26: number analyzed (Participants) | 174 | 173
  Communication, CFB to Week 26 | -2.4 (0.21) | -2.0 (0.19)
  Emotion/affect, BL: number analyzed (Participants) | 198 | 200
  Emotion/affect, BL | 12.7 (0.14) | 12.5 (0.15)
  Emotion/affect, CFB to Week 26: number analyzed (Participants) | 171 | 172
  Emotion/affect, CFB to Week 26 | -1.9 (0.17) | -1.6 (0.15)
  Social Involvement, BL: number analyzed (Participants) | 198 | 199
  Social Involvement, BL | 13.1 (0.16) | 12.6 (0.18)
  Social Involvement, CFB to Week 26: number analyzed (Participants) | 173 | 172
  Social Involvement, CFB to Week 26 | -2.0 (0.17) | -1.4 (0.19)
  Motivation, BL: number analyzed (Participants) | 198 | 201
  Motivation, BL | 16.7 (0.18) | 16.6 (0.18)
  Motivation, CFB to Week 26: number analyzed (Participants) | 173 | 173
  Motivation, CFB to Week 26 | -2.6 (0.20) | -2.2 (0.23)
  Retardation, BL | 7.0 (0.12) | 7.0 (0.12)
  Retardation, CFB to Week 26: number analyzed (Participants) | 174 | 173
  Retardation, CFB to Week 26 | -1.7 (0.13) | -1.5 (0.13)

6. Secondary Outcome: Change From Baseline to Week 26 in the Clinical Global Impression of Schizophrenia Scale-Severity (CGI-SCH-S) of Negative Symptoms Score
Description: The CGI-SCH-S is a clinician-rated, 7-point scale to evaluate positive, negative, depressive, cognitive symptoms and overall severity in schizophrenia. For the purpose of this study, only the negative symptoms were evaluated. The score could range from 1 (normal, not ill) to 7 (among the most severely ill).
Time Frame: From baseline to Week 26
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Pimavanserin | Placebo
Number analyzed (Participants) | 199 | 201
score on a scale
  Baseline | 4.6 (0.04) | 4.7 (0.04)
  Change from baseline to Week 26: number analyzed (Participants) | 174 | 173
  Change from baseline to Week 26 | -0.6 (0.06) | -0.6 (0.06)

7. Secondary Outcome: Clinical Global Impression of Schizophrenia Scale-Improvement (CGI-SCH-I) of Negative Symptoms Score at Week 26
Description: The CGI-SCH-I is a clinician-rated, 7-point scale to evaluate change from baseline in positive, negative, depressive, cognitive symptoms and overall severity in schizophrenia. For the purpose of this study, only the changes in negative symptoms from baseline were evaluated. The score could range from 1 (very much improved) to 7 (very much worse).
Time Frame: From baseline to Week 26
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Pimavanserin | Placebo
Number analyzed (Participants) | 174 | 173
score on a scale | 3.1 (0.07) | 3.1 (0.06)

8. Secondary Outcome: Proportion of CGI-SCH-I Responders (CGI-SCH-I Score of 1 or 2) at Week 26; Observed Cases
Description: The CGI-SCH-I is a clinician-rated, 7-point scale that is designed to evaluate change from baseline in positive, negative, depressive, cognitive symptoms and overall severity in schizophrenia. For the purpose of this study, only the changes in negative symptoms from baseline were evaluated. The 7-point scores range from 1 (very much improved) to 7 (very much worse); responders were defined as those with CGI-SCH-I of 1 or 2.
  The analysis includes observed cases; missing cases were not imputed.
Time Frame: From baseline to Week 26
Population: Patients who were randomised and treated (received at least one dose of study drug); had a baseline value and at least one post-baseline value for NSA-16 total score; and had no missing values at Week 26.
Measure: Count of Participants; unit: Participants
Arm/Group | Pimavanserin | Placebo
Number analyzed (Participants) | 174 | 173
Participants | 47 | 40

9. Secondary Outcome: Change From Baseline to Week 26 in the Positive and Negative Syndrome Scale (PANSS) Total Score
Description: The PANSS is a 30-item scale to evaluate the presence, absence, and severity of schizophrenia symptoms. Items are scored over the past week (7 days) on a 7-point scale from 1 (absent) to 7 (extreme). The PANSS total score is the sum of scores and ranges from a minimum of 30 to a maximum of 210. Higher scores denote more severe symptoms.
Time Frame: From baseline to Week 26
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Pimavanserin | Placebo
Number analyzed (Participants) | 199 | 201
score on a scale
  Baseline | 77.2 (0.70) | 79.4 (0.62)
  Change from baseline to Week 26: number analyzed (Participants) | 174 | 173
  Change from baseline to Week 26 | -8.7 (0.75) | -8.6 (0.76)

10. Secondary Outcome: Change From Baseline (CFB) to Week 26 in PANSS Subscale Scores
Description: The PANSS is a 30-item scale to evaluate the presence, absence, and severity of schizophrenia symptoms. Items are scored over the past week (7 days) on a 7-point scale from 1 (absent) to 7 (extreme). The PANSS has 3 subscales that are the sums of the respective item scores, including the positive scale (min 7, max 49), negative scale (min 7, max 49), and general psychopathology scale (min 16, max 112). Higher scores denote more severe symptoms.
Time Frame: From baseline (BL) to Week 26
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Pimavanserin | Placebo
Number analyzed (Participants) | 199 | 201
score on a scale
  Positive subscale, BL | 13.1 (0.24) | 13.7 (0.22)
  Positive subscale, CFB to Week 26: number analyzed (Participants) | 174 | 173
  Positive subscale, CFB to Week 26 | -0.6 (0.19) | -0.8 (0.21)
  Negative subscale, BL | 27.5 (0.26) | 27.5 (0.25)
  Negative subscale, CFB to Week 26: number analyzed (Participants) | 174 | 173
  Negative subscale, CFB to Week 26 | -4.0 (0.29) | -3.8 (0.31)
  General psychopathology subscale, BL | 36.6 (0.44) | 38.2 (0.40)
  General psychopathology subscale, CFB to Week 26: number analyzed (Participants) | 174 | 173
  General psychopathology subscale, CFB to Week 26 | -4.1 (0.43) | -4.0 (0.43)

11. Secondary Outcome: Change From Baseline to Week 26 in Brief Assessment of Cognition in Schizophrenia (BACS) Composite Score
Description: The BACS is a performance-based assessment of treatment-related changes in cognition, assessing 6 domains of verbal memory and learning; working memory; motor function; verbal fluency; attention and speed of processing; and executive function. The 6 domains with their raw scores are: verbal memory 0-75; digit sequencing 0-28; token motor 0-100; verbal fluency 0-225; symbol coding 0-110; Tower of London 0-22. For each domain, higher scores reflect better cognition. Raw scores are converted to age and sex-corrected normalized scores. The BACS composite score is calculated as the mean of the normalized scores from the 6 subscale scores, standardized so that the mean of the BACS composite score in the healthy normative sample is 50 and the standard deviation is 10.
Time Frame: From baseline to Week 26
Population: Patients who were randomised and treated (received at least one dose of study drug) and had a baseline value and at least one post-baseline value for NSA-16 total score. Analysis only included patients with data/endpoint assessment and additionally excluded patients with raw scores outside of the score range.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Pimavanserin | Placebo
Number analyzed (Participants) | 197 | 199
score on a scale
  Baseline | 22.94 (1.271) | 20.99 (1.198)
  Change from baseline to Week 26: number analyzed (Participants) | 173 | 170
  Change from baseline to Week 26 | 3.33 (0.719) | 4.16 (0.696)

12. Secondary Outcome: Change From Baseline to Week 26 in 10-item Drug Attitude Inventory (DAI-10) Score
Description: The DAI-10 contains 6 items (1, 3, 4, 7, 9, and 10) that a subject who is fully adherent to the prescribed medication would answer as "True" and 4 items (2, 5, 6, and 8) that a subject who is fully adherent to the prescribed medication would answer as "False." A correct answer is scored +1 and an incorrect answer is scored -1. The total score is the sum of pluses and minuses, which can range from -10 to 10 in increments of 2. A positive total score indicates a positive subjective response (adherent) and a negative total score indicates a negative subjective response (non-adherent). Higher scores denote better adherence.
Time Frame: From baseline to Week 26
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Pimavanserin | Placebo
Number analyzed (Participants) | 199 | 201
score on a scale
  Baseline | 5.7 (0.22) | 5.7 (0.23)
  Change from baseline to Week 26: number analyzed (Participants) | 174 | 173
  Change from baseline to Week 26 | 0.2 (0.23) | 0.2 (0.19)

13. Secondary Outcome: Change From Baseline to Week 26 in Karolinska Sleepiness Scale (KSS) Score
Description: The KSS is a self-reported subjective measure of a subject's level of drowsiness. Respondents must choose statements that most accurately describe their level of sleepiness over the past 7 days. Scoring was based on a 9-point verbally anchored scale ranging from 1 (extremely alert) to 9 (very sleepy, great effort to keep awake, fighting sleep). Higher scores denoted more drowsiness.
Time Frame: From baseline to Week 26
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Pimavanserin | Placebo
Number analyzed (Participants) | 199 | 201
score on a scale
  Baseline | 4.6 (0.11) | 4.8 (0.10)
  Change from baseline to Week 26: number analyzed (Participants) | 174 | 173
  Change from baseline to Week 26 | -0.3 (0.12) | -0.6 (0.13)

ADVERSE EVENTS:
Time Frame: From the time of the first dose of study drug until 30 days after the last dose of study drug planned to be administered at Week 26
Description: The analysis population were all patients randomised and treated (i.e. receiving at least one dose of study drug).
Arm/Group | Pimavanserin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/201 | 0/202
Serious Adverse Events (participants affected / at risk) | 4/201 | 1/202
Other Adverse Events (participants affected / at risk) | 20/201 | 19/202
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pimavanserin (N=201) | Placebo (N=202)
Schizophrenia (Psychiatric disorders) | 4 (4) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pimavanserin (N=201) | Placebo (N=202)
Headache (Nervous system disorders) | 13 (17) | 10 (10)
Somnolence (Nervous system disorders) | 11 (12) | 10 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator may publish the study results, relative to his/her own patients, only after review, comment and approval by the sponsor. No publication of confidential information shall be made without the sponsor's Prior written consent. At least 60 days prior to submitting a manuscript or prior to any public presentation, a copy of the manuscript or presentation will be provided to the sponsor for review and comment. The sponsor has 60 days to review and comment

DOCUMENTS (2):
  • Study Protocol (2017-03-31): https://cdn.clinicaltrials.gov/large-docs/05/NCT02970305/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-01): https://cdn.clinicaltrials.gov/large-docs/05/NCT02970305/SAP_001.pdf